CLINICAL TRIAL: NCT06542263
Title: Clinical Study on the Effect of Continuous Positive Airway Pressure Ventilation on Atrial Fibrillation Recurrence After Catheter Ablation in Patients with Atrial Fibrillation and Obstructive Sleep Apnea
Brief Title: Clinical Study on the Effect of CPAP on AF Recurrence After Catheter Ablation in Patients with AF and OSA
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-LK2024034-IR01
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Continuous Positive Airway Pressure; Obstructive Sleep Apnea; Recurrence; Observational Study
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- non-CPAP group: The non-CPAP group underwent catheter ablation and conventional treatment for AF combined with OSA
  Interventions: Device: CPAP
- CPAP group: The CPAP group underwent catheter ablation and CPAP treatment for AF combined with OSA

INTERVENTIONS:
Device: CPAP — For the non-CPAP group, the intervention includes catheter ablation and conventional treatment for AF combined with OSA; For the CPAP group, the intervention includes catheter ablation and CPAP treatment for AF combined with OSA
  Groups: non-CPAP group

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia in clinical practice, significantly increasing the risks of death, stroke, heart failure, cognitive impairment, and dementia, thus severely impacting patients' quality of life. However, for AF patients with concomitant cardiovascular risk factors, particularly those with obstructive sleep apnea (OSA), the success rate of catheter ablation is significantly reduced. Continuous positive airway pressure (CPAP) is currently an effective treatment for OSA, effectively correcting nocturnal intermittent hypoxia and fragmented sleep caused by OSA. However, the effect of CPAP therapy on AF recurrence in patients with OSA undergoing catheter ablation remains controversial. Faced with conflicting research findings, our team recently conducted a meta-analysis (registration number CRD42023398588) to assess the impact of CPAP on AF recurrence post catheter ablation in patients with AF and OSA, suggesting that CPAP significantly reduces AF recurrence post catheter ablation (RR = 0.58, P < 0.01). However, considering the limited number of included studies, potential bias risks, and confounding factors, our meta-analysis results await further confirmation through real-world studies by our team. Therefore, our team plans to conduct further research on the impact of CPAP on AF recurrence post catheter ablation in patients with moderate to severe OSA, aiming to provide clinical guidance for the treatment of AF in patients with moderate to severe OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of AF combined with moderate to severe OSA (OSA diagnostic criteria: apnea hypopnea index (AHI) greater than 15/hour, and at least 80% of all events are respiratory sleep obstructive events; AF includes persistent atrial fibrillation and paroxysmal atrial fibrillation)
2. Age ≥ 18 years old
3. The patient voluntarily participates in the project and signs informed consent
4. All patients undergo overnight sleep pressure titration at the sleep center to determine the minimum pressure value for continuous positive airway pressure ventilation at home. All patients are required to undergo CPAP treatment at home at least 5 days a week, with each session lasting at least 4 hours

Exclusion Criteria:

1. Patients with neuromuscular disorders, pulmonary hypopnea, and severe lung diseases
2. Preoperative confirmation of thrombus in the left atrium
3. The patient has no desire for conversion
4. Secondary atrial fibrillation (hyperthyroidism, tumors, etc.)
5. Individuals with contraindications to anticoagulants
6. Left atrial diameter (LAD) exceeding 60mm (2D echocardiography long axis section data)
7. Pregnant women
8. History of myocardial infarction, percutaneous coronary intervention, and cardiac surgery in the past three months
9. Stroke or transient ischemic attack in the past six months
10. After artificial valve implantation surgery
11. Severe renal insufficiency (creatinine Cr>2.5mg/dl or>221umol/L, or glomerular filtration rate eGFR<30ml/min/1.73m2)
12. Acute diseases or active infections that occur before surgery, recorded as pain, fever, positive blood culture, and/or leukocytosis, or have been treated with antibiotics.
13. Expected survival period<1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of AF combined with moderate to severe OSA (OSA diagnostic criteria: apnea hypopnea index (AHI) greater than 15/hour, and at least 80% of all events are respiratory sleep obstructive events; AF includes persistent atrial fibrillation and paroxysmal atrial fibrillation)
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
AF recurrence after ablation | At 3, 6, 9, and 12 months after AF ablation
  AF recurrence after ablation via Surface electrocardiogram and 24-hour dynamic electrocardiogram examination. If there are symptoms, seek medical attention at any time for electrocardiogram examination
AF burden after ablation AF burden after ablation AF burden after ablation | At 3, 6, 9, and 12 months after AF ablation
  AF burden after ablation via 24-hour dynamic electrocardiogram examination AF burden after ablation via 24-hour dynamic electrocardiogram examinatio AF burden after ablation via 24-hour dynamic electrocardiogram examinatio

SECONDARY OUTCOMES:
The recurrence of AF after combination with antiarrhythmic drugs | At 3, 6, 9, and 12 months after AF ablation
  The recurrence of AF after combination with antiarrhythmic drugs via Surface electrocardiogram and 24-hour dynamic electrocardiogram examination. If there are symptoms, seek medical attention at any time for electrocardiogram examination
AF burden after combination with antiarrhythmic drugs | At 3, 6, 9, and 12 months after AF ablation
  AF burden after combination with antiarrhythmic drugs via 24-hour dynamic electrocardiogram examinatio
SF-36 | At 3 and 12 months after AF ablation
  SF-36 with standard scores ranging from 0 to 100. The higher the score, the better the health status
Euro-QoL5D Survey Scoring | At 3 and 12 months after AF ablation
  Euro-QoL5D survey questionnaire is between 0 and 100, with higher scores indicating better health status

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jinagsu, China

IPD SHARING:
Plan to Share IPD: Undecided